CLINICAL TRIAL: NCT03253783
Title: The Evaluation of Pulse: A Mobile Health App and Teen Pregnancy Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy Teen Network (Other)
Collaborators: Child Trends (Other); Ewald and Wasserman (Unknown); Meta Media (Unknown)
Responsible Party: Principal Investigator, Martinez Garcia, Dr. Genevieve Martínez-García, Healthy Teen Network
Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000038
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Unprotected Sex; Contraceptive Usage; Reproductive and Sexual Health Care Utilization
MeSH Terms: conditions — Unsafe Sex; Contraception Behavior | interventions — Pulse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Pulse

SUMMARY:
This study uses a randomized controlled design to evaluate the efficacy of a new mobile app, Pulse, in reducing the incidence of unprotected sex among young women. Pulse is a web-based mobile health application that can be accessed through mobile smartphones and computers. Pulse was designed to increase highly effective birth control use and reproductive and sexual health care utilization, and ultimately decrease teen pregnancy. The sample is comprised of women with the following characteristics at study enrollment: aged 18-20, not pregnant or trying to become pregnant, has daily access to a smartphone, currently living in the United States or a U.S. territory, and speaks either English or Spanish. Most of the sample (at least 70%) will be women who identify as Black and/or Latina. The evaluation team plans to enroll up to 1,300 participants over a one-year enrollment period using social media, including Facebook, Instagram, and Twitter.

Users access Pulse autonomously, on their own terms, and in their own time and place. The app consists of 6 sections and includes 3 hours of unique content. It does not require the user to follow a specific sequence of content viewed; however, all users will receive a monetary incentive after registering with the apps. Youth randomized to the intervention condition are given access to Pulse indefinitely and receive daily text messages related to sexual health for 6 weeks. Control participants are directed to a free general health/fitness web-based mobile application, also called Pulse, and receive text messages related to general health for 6 weeks. The control and treatment apps look and feel similar aesthetically but contain different content. Participants in both the intervention and comparison groups receive a baseline survey and a 6-week follow-up survey. Participants will also receive incentives once they complete the baseline and post-intervention survey. Both surveys are conducted online via an electronic survey platform. This study is being conducted as a Rigorous Evaluation of New or Innovative Approaches to Prevent Teen Pregnancy funded by the U.S. Department of Health and Human Services' Office of Adolescent Health.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* Age Limit: 18-20
* Must have daily access to a smartphone that receives text messages and can access to the Internet
* Must speak English or Spanish
* Must live in the United States or a U.S. territory

Exclusion Criteria:

* Currently pregnant or trying to get pregnant

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1304 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Unprotected sex, no contraceptive | 6-week post-baseline (in the past 6 weeks)
  Ever having sexual intercourse without using any method of contraception (among full sample)
Unprotected sex, no highly effective contraceptive | 6-week post-baseline (in the past 6 weeks)
  Ever having sexual intercourse without using a hormonal or LARC method of contraception (among full sample)

SECONDARY OUTCOMES:
Reproductive and sexual health care utilization (among full sample) | 6-weeks post-baseline
  Visiting a health care provider for reproductive or sexual health services within the past 6 weeks for the 1st follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Martinez-Garcia, PhD, Principal Investigator — Healthy Teen Network; Jennifer Manlove, PhD, Principal Investigator — Child Trends
Locations (1):
- Healthy Teen Network, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730